CLINICAL TRIAL: NCT00633932
Title: A Multicentre, Randomised, Double-blind, Parallel-group, Comparative Study to Compare the Efficacy and Safety of Esomeprazole 20 mg and 40 mg Once Daily Oral Administration With Omeprazole 20 mg Once Daily Oral Administration in Patients With Reflux Esophagitis
Brief Title: Reflux Esophagitis Phase III Study (Initial Treatment)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind / Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D961HC00002
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Results first posted 2010-04-08 (Estimated); Last update posted 2010-12-20 (Estimated); Status verified 2010-12

CONDITIONS: Reflux Esophagitis
Keywords: Reflux Esophagitis
MeSH Terms: conditions — Esophagitis, Peptic | interventions — Esomeprazole; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Esomeprazole 20mg
  Interventions: Drug: Esomeprazole
- 2 (Experimental): Esomeprazole 40mg
  Interventions: Drug: Esomeprazole
- 3 (Active Comparator): Omeprazole 20mg
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Esomeprazole — 20mg once daily
  Other Names: Nexium
  Arms: 1
Drug: Esomeprazole — 40 mg once daily
  Other Names: Nexium
  Arms: 2
Drug: Omeprazole — 20mg once daily
  Other Names: Prilosec
  Arms: 3

SUMMARY:
This study is to evaluate the efficacy of esomeprazole 20 mg once daily and 40 mg once daily for 8 weeks on healing of Reflux Esophagitis in patients with reflux esophagitis in comparison with omeprazole 20 mg once daily by assessment of presence/absence of Reflux Esophagitis at Week 8 according to the Los Angeles classification .

ELIGIBILITY:
Inclusion Criteria:

* Endoscopically verified Reflux Esophagitis classified into Los Angeles classification Grade A, B, C or D within 1 week before randomisation

Exclusion Criteria:

* Gastric or duodenal ulcer verified by EGD within 12 weeks before randomisation.
* Use of any PPI from 14 days before EGD performed at the screening visit to the day of randomisation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2007-12; Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maotsugu Oyama, MD, PhD, Study Director — AstraZeneca
Locations (41):
- Japan (41):
  - Research Site, Akita, Akita
  - Research Site, Kashiwa, Chiba
  - Research Site, Kisarazu, Chiba
  - Research Site, Kōriyama, Fukishima
  - Research Site, Nihonmatsu, Fukishima
  - Research Site, Nishishirakawa, Fukishima
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kurume, Fukuoka
  - Research Site, Nukaya, Fukuoka
  - Research Site, Shirakawa, Fukushima
  - Research Site, Sugawa, Fukushima
  - Research Site, Gifu, Gifu
  - Research Site, Maebashi, Gunma
  - Research Site, Yasunaka, Gunma
  - Research Site, Sapporo, Hokkaido
  - Research Site, Hitachi, Ibaraki
  - Research Site, Mito, Ibaraki
  - Research Site, Tsukuba, Ibaraki
  - Research Site, Sakaidechō, Kagawa-ken
  - Research Site, Takamatsu, Kagawa-ken
  - Research Site, Fujisawa, Kanagawa
  - Research Site, Kawasaki, Kanagawa
  - Research Site, Sagamihara, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kyoto, Kyoto
  - Research Site, Shibata, Myagi
  - Research Site, Kiso, Nagano
  - Research Site, Matsumoto, Nagano
  - Research Site, Ōita, Oita Prefecture
  - Research Site, Fujiidera, Osaka
  - Research Site, Toyonaka, Osaka
  - Research Site, Shizuoka, Shizuoka
  - Research Site, Ohtawara, Tochigi
  - Research Site, Toshima-ku, Tokayo
  - Research Site, Adachi City, Tokyo
  - Research Site, Hachiōji, Tokyo
  - Research Site, Kiyose, Tokyo
  - Research Site, Setagaya City, Tokyo
  - Research Site, Shinagawa, Tokyo
  - Research Site, Tottori-shi, Tottori
  - Research Site, Shimonoseki, Yamaguchi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled on 11 December 2007. Last subject completed on 12 December 2008.
Pre-assignment Details: Out of 602 enrolled subjects, 572 subjects were randomised and 30 subjects were not randomised. The reasons of no randomisation were 'Incorrect enrollment' (25 subjects) and 'Voluntary discontinuation by Subject' (5 subjects).
Groups:
- Experimental: Esomeprazole 40mg: Esomeprazole 40mg once daily
- Experimental: Esomeprazole 20mg: Esomeprazole 20mg once daily
- Comparator: Omeprazole 20mg: Omeprazole 20mg once daily
Period: Overall Study
Arm/Group | Experimental: Esomeprazole 40mg | Experimental: Esomeprazole 20mg | Comparator: Omeprazole 20mg
Started | 191 (Randomised) | 190 (Randomised) | 191 (Randomised)
Completed | 179 | 176 | 180
Not Completed | 12 | 14 | 11
Not completed — Adverse Event | 1 | 3 | 4
Not completed — Withdrawal by Subject | 3 | 9 | 1
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Protocol Violation | 5 | 2 | 3
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Doctor's judgement | 1 | 0 | 0
Not completed — Moved Away | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Esomeprazole 40mg | Experimental: Esomeprazole 20mg | Comparator: Omeprazole 20mg | Total
Number analyzed (Participants) | 191 | 190 | 191 | 572
Age, Customized [Number; unit: Participants]
  < 65 years | 127 | 135 | 126 | 388
  65 - 74 years | 47 | 36 | 44 | 127
  >= 75 years | 16 | 18 | 20 | 54
  Missing | 1 | 1 | 1 | 3
Sex/Gender, Customized [Number; unit: Participants]
  Male | 139 | 137 | 134 | 410
  Female | 51 | 52 | 56 | 159
  Missing | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Healing of Reflux Esophagitis (RE) Who Were Graded "O" at Week 8 Out of Patients Who Were Graded "A, B, C or D" at Baseline According to Los Angeles Classification".
Description: Los Angeles classification consists of 5 grades (Grade O, Grade A, Grade B, Grade C, Grade D). The subjects who were definitely diagnosed to have RE classified into LA classification Grade A, B, C or D based on the EGD on Visit 1 were randomised. A subject classified into LA classification Grade O was considered no reflux esophagitis. The definitions of each grade are: Grade A (Mucosal break < 5 mm in length), Grade B (Mucosal break > 5mm), Grade C (Mucosal break continuous between > 2 mucosal folds) and Grade D (Mucosal break >75% of esophageal circumference).
Time Frame: 8 weeks
Population: One participant for each treatment group did not take any investigational product. These 3 participants were excluded (1 for each treatment group) from all the efficacy and safety analyses.
Measure: Number; unit: participants
Arm/Group | Experimental: Esomeprazole 40mg | Experimental: Esomeprazole 20mg | Comparator: Omeprazole 20mg
Number analyzed (Participants) | 190 | 189 | 190
participants | 171 | 165 | 166

2. Secondary Outcome: Number of Participants With Healing of Reflux Esophagitis (RE) Who Were Graded "O" at Week 4 Out of Patients Who Were Graded "A, B, C or D" at Baseline According to Los Angeles Classification
Description: Los Angeles classification consists of 5 grades (Grade O, Grade A, Grade B, Grade C and Grade D). The subjects who were definitely diagnosed to have RE classified into LA classification Grade A, B, C or D based on the EGD on Visit 1 were randomised. A subject classified into LA classification Grade O was considered no reflux esophagitis. The definitions of each grade are: Grade A (Mucosal break < 5 mm in length), Grade B (Mucosal break > 5mm), Grade C (Mucosal break continuous between > 2 mucosal folds) and Grade D (Mucosal break >75% of esophageal circumference).
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Experimental: Esomeprazole 40mg | Experimental: Esomeprazole 20mg | Comparator: Omeprazole 20mg
Number analyzed (Participants) | 190 | 189 | 190
participants | 141 | 147 | 143

ADVERSE EVENTS:
Description: One patient for each treatment group did not take any investigational product.
Arm/Group | Experimental: Esomeprazole 40mg | Experimental: Esomeprazole 20mg | Comparator: Omeprazole 20mg
Serious Adverse Events (participants affected / at risk) | 0/190 | 1/189 | 1/190
Other Adverse Events (participants affected / at risk) | 12/190 | 9/189 | 16/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Esomeprazole 40mg (N=190) | Experimental: Esomeprazole 20mg (N=189) | Comparator: Omeprazole 20mg (N=190)
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Influenza Like Illness (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Esomeprazole 40mg (N=190) | Experimental: Esomeprazole 20mg (N=189) | Comparator: Omeprazole 20mg (N=190)
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 6
Nasopharyngitis (Infections and infestations) | 10 | 6 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs were prohibited to disclose all information related to this study withiout AZ approval before this study was completed.